CLINICAL TRIAL: NCT03171155
Title: Prospective, Multi-Center, Single Arm Study of the Medeon Biodesign XPro™ Suture-Mediated Vascular Closure Device System
Brief Title: Clinical Study of the Medeon Biodesign XPro™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medeon Biodesign, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-LHC03
Record Dates: First submitted 2017-05-23; First posted 2017-05-31 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Percutaneous Closure of Arteriotomy in Common Femoral Artery

STUDY DESIGN:
Intervention Model Description: Implantation of the XPro System
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- XPro System (Experimental): Implantation of XPro System during percutaneous vascular closure
  Interventions: Device: XPro System

INTERVENTIONS:
Device: XPro System — Implantation of the XPro System

SUMMARY:
To access the safety and performance of the XPro System to facilitate hemostasis in patients undergoing percutaneous endovascular procedures utilizing 8-18 Fr introducer sheath via the common femoral.

DETAILED DESCRIPTION:
This is a prospective multi-center, single arm study to assess the safety and performance of the XPro System compared to a historical control developed from published studies of two marketed competitive devices, Perclose ProGlide® and Prostar® XL (both from Abbott Vascular, Inc., Redwood City, CA, USA). The goal of the study is to show that XPro System is non-inferior to the competitors in efficacy and safety. Patients scheduled for percutaneous BAV, TAVR/TAVI, EVAR, or TEVAR procedures using an 8-18 Fr introducer sheath will be screened for study eligibility. Patients will be followed for 30 days post procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient is > 18 years old
* Patient is scheduled for percutaneous BAV, TAVR/TAVI, EVAR, or TEVAR involving access through the femoral artery using an 8-18 Fr introducer sheath
* Patient is able to undergo emergent vascular surgery if a complication related to the vascular closure necessitates such surgery
* Patient, or authorized representative, signs a written Informed Consent form to participate in the study, prior to any study mandated procedures
* Patient is willing and able to complete follow-up

Exclusion Criteria:

* Prior intra-aortic balloon pump at access site
* Patients with severe claudication, iliac or femoral artery diameter stenosis greater than 50%
* Common femoral artery lumen diameter is < 6 mm
* Prior target artery closure with any closure device < 90 days, or closure with manual compression ≤ 30 days prior to index procedure
* Prior vascular surgery, vascular graft, or stent in region of access site
* Patients receiving glycoprotein IIb/IIIa inhibitors before, during, or after the catheterization procedure
* Patients with significant anemia ((Hgb < 10 g/dL, Hct < 30%)
* Patient with known bleeding disorder including thrombocytopenia (platelet count < 100,000), thrombasthenia, hemophilia or Von Willebrand's disease
* Patients with renal insufficiency (serum creatinine level > 221µmol/L) or renal transplant
* Known allergy to contrast reagent
* Inability to tolerate aspirin and/or other anticoagulation treatment
* Planned anticoagulation therapy post-procedure such that ACT is expected to be elevated above 350 seconds for more than 24 hours after the procedure
* Connective tissue disease (e.g., Marfan's Syndrome)
* Thrombolytics (e.g. t-PA, streptokinase, urokinase), Angiomax (bivalirudin) or other thrombin-specific anticoagulants ≤ 24 hours prior to the procedure
* Recent (within 8 weeks) cerebrovascular accident or Q-wave myocardial infarction
* Patients who are morbidly obese BMI > 40 kg/m2
* Planned major intervention or surgery within 30 days following the interventional procedure
* Patients who are unable to ambulate at baseline
* Currently participating in a clinical study of an investigational device or drug that has not completed study endpoint
* Known allergy to any device component
* Patient is known or suspected to be pregnant or lactating
* Life expectancy < 1 year as judged by the investigator
* Patient has other medical, social or psychological problem that in the opinion of the investigator precludes them from participating Intra-Procedure
* Access site above the most inferior border of the inferior epigastric artery (IEA) and/or above the inguinal ligament based upon bony landmarks
* Access site in the profunda femoris or superficial femoral arteries, or the bifurcation of these vessels
* Ipsilateral femoral venous sheath during the catheterization procedure
* Common femoral artery calcium, which is fluoroscopically visible
* Patients where there is difficulty inserting the introducer sheath or greater than 2 ipsilateral arterial punctures at the start of the catheterization procedure
* Difficulty in obtaining vascular access resulting in multiple arterial punctures and/or posterior arterial puncture
* Evidence of a pre-existing hematoma, arteriovenous fistula, or pseudoaneurysm at the access site
* Patients with intra-procedural bleeding around access site
* Evidence of active systemic or local groin infection
* Patients receiving glycoprotein IIb/IIIa inhibitors during, or after the catheterization procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Time to Hemostasis | 15 minutes
  Time to hemostasis absent of any access-site-related adjunctive surgical or endovascular procedures.
Freedom from major VARC-2 events | Up to 30 days of procedure
  Freedom from major VARC-2 events within 30 days of the procedure.

SECONDARY OUTCOMES:
Freedom from minor VARC-2 events | Up to 30 days of procedure
  Freedom from minor VARC-2 events up to 30 days of the procedure.
Successful hemostasis with the XPro System | at 48 hours or at discharge from hospital, whichever comes first; and up to 30 days post-procedure
  Without the need for any access-site-related adjunctive surgical or endovascular procedures and freedom from major VARC-2 events.
Freedom from access-site infection | Up to 30 days of procedure
  Freedom from access-site infection requiring IV or IM antibiotics, or extended hospitalization or re-hospitalization.

OTHER OUTCOMES:
Time to ambulation | Up to 48 hours
  Defined as elapsed time from sheath removal and time when the patient stands and walks at least 20 feet without re-bleeding.
Time to hospital discharge | Up to 2 weeks
  Time to actual hospital discharge defined as elapsed time from sheath removal to actual physical discharge from the hospital.

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (2):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - St. Vincent's Hospital Melbourne, Fitzroy, Victoria
- New Zealand (3):
  - Auckland City Hospital, Auckland
  - Christchurch Hosptial, Christchurch
  - Waikato Hospital, Hamilton
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No